CLINICAL TRIAL: NCT01672372
Title: The Effect of Methylated Vitamin B Complex on Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Premier Research Labs (Other)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20091119
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Max Stress B (Placebo Comparator): oil/water emulsion with food coloring to simulate actual product
  Interventions: Dietary Supplement: Placebo Max Stress B
- Max Stress B (Experimental): whole-nutrient natural source extract from probiotic colonies that contains vitamins B1, B2, B5, B6, B12, and folate, PABA, biotin, inositol, purified water and certified organic alcohol.
  Interventions: Dietary Supplement: Max Stress B

INTERVENTIONS:
Dietary Supplement: Max Stress B — Participants are to mix one vial per day of either placebo or actual supplement in 1 liter of water and drink over the course of the day
  Arms: Max Stress B
Dietary Supplement: Placebo Max Stress B
  Arms: Placebo Max Stress B

SUMMARY:
The proposed study is a 60-day, randomized, double-blind, placebo-controlled trial to evaluate the efficacy of a methylated vitamin B complex nutritional supplement (Max Stress B™) for improving depressive and anxiety symptoms according to the Beck Depression and Anxiety Inventories, respectively, in 60 patients (18+ years of age) diagnosed with major depression or other forms of depressive disorders and an elevated level of homocysteine (> 10 µmol/L) at baseline. Secondary outcomes will include anthropometrics for body composition, blood pressure and pulse, level of physical activity, dietary intake, and quality of life. Participants will be assessed at baseline and 30 and 60 days. The study will consist of two treatment arms: (a) vitamin B complex nutritional supplement and (b) placebo.

The information obtained in this study will help in determining the efficacy of using nutritional supplements for improving the outcomes of people with depression.

DETAILED DESCRIPTION:
Study Design Potential participants will be identified through referrals from the offices of Dr. Woolger, the UM Department of Psychiatry Clinics, the Medical Wellness Center, and the Center for Complementary and Integrative Medicine. Drs. Woolger and Konefal will conduct a preliminary screening of their clients to determine if the potential participant meets the inclusion criteria to participate in the study. Dr. Lewis, Messrs. Long, Dicenso, or Bregman, or Mses. Hoffman, Rafatjah, Melillo, Ko, Alonso, or McCurdy will conduct preliminary screenings through the Medical Wellness Center or the Center for Complementary and Integrative Medicine. Once accepted into the study, participants will then contact Dr. Lewis, Messrs. Long, Dicenso, or Bregman, or Mses. Hoffman, Rafatjah, Melillo, Ko, Alonso, or McCurdy for informed consent and study protocol procedures. Subjects will then be assigned to one of the two study conditions. Assignment of subjects to treatment groups will be done by following a table of random permutations, which will balance the number of subjects in each group. The table will be prepared in advance by a random number generating program.

Participants Sixty subjects (30 in each condition) with depression will participate in this study. Subjects will be primarily those who have expressed an interest in trying non-medication or integrative treatment approaches for their depression.

Initial visit The study will be fully explained to each potential participant, and a written informed consent will be obtained before beginning the intervention. Dr. Lewis, Messrs. Long, Dicenso, or Bregman, or Mses. Hoffman, Rafatjah, Melillo, Ko, Alonso, or McCurdy will administer all of the assessments at baseline and follow-up and will notify the subjects of the time to return for the follow-up appointments.

Intervention Participants enrolled in the study will receive either the Max Stress B™ at a dosage level of ½ teaspoon twice daily or the placebo for the 60-day treatment period. Subjects will not be advised to modify eating or physical activity habits or non-depression prescription medication use. Subjects will not be allowed to use depression-treatment medication starting at 2 weeks before beginning the intervention and until the conclusion of the 60-day treatment period. Subjects will be instructed not to consume any other nutritional supplements containing any of the vitamin B complex nutrients, SAMe, inositol, PABA, or folate for two weeks prior to having the baseline assessments and until the conclusion of the 60-day period. Because of how Max Stress B™ is produced by Premier Research Labs, consuming the Max Stress B™ should be well-tolerated. We are aware of no side effects of this particular product. According to the company's literature, Max Stress B™ is a whole-nutrient natural source extract from probiotic colonies that contains: vitamins B1, B2, B3, B5, B6, and B12, and folate, PABA, biotin, inositol, purified water, and certified organic alcohol. This product is documented online at the following web address: http://www.prlabs.com/ under the "Products" tab, item #2352.

Outcomes and Assessments Each participant will complete a basic demographics and medical history questionnaire to assess the importance of these background variables. They will also be asked to list their current medications and note any changes in type or amount during the course of the study. Blood pressure, heart rate, body weight and height, skinfold assessments, and hip and waist circumference will be assessed by Dr. Lewis, Messrs. Long, Dicenso, Bregman, or Reihm, or Mses. Rafatjah, Melillo, Ko, Alonso, or McCurdy at baseline and 30- and 60-days follow-up.

Criteria used to select the assessment instruments included: a) appropriateness for the population; b) ease of administration and scoring; c) experience administering these measures; and d) employment of measures involving a multi-method (i.e., self-report and physical measures) approach to enhance the validity of the overall assessment.

The following measures will be assessed:

1. The primary outcome of this study is depression level, assessed by the Beck Depression Inventory II, which will be assessed to reflect its relationship to changes in dietary patterns and physical activity. Because item 9 of the Beck Depression Inventory inquires about "Suicidal thoughts or wishes," we will immediately notify the attending physician in the Crisis facility of UM/JMH if a subject responds affirmatively to this question, which may be indicative of suicidal ideation (SI). Any spontaneous comments or circumstances indicative of SI should be explored with the participant (e.g., "life not worth living," "be better off dead," selling or giving away possessions, or withdrawing from relationships, etc.). If suicidal ideation is present, the assessor will maintain persistent contact with the subject until the physician can meet with the subject. If the suicide threat is judged to be immediate by the physician (i.e., the subject indicates current intent, has a plan, and available means) then the assessor will maintain contact with the subject and ensure that the subject is taken to a psychiatric emergency setting. The Jackson Crisis Mental Health Unit (305-355-7777) is a potential emergency facility and is located at 1695 N.W. 9th Avenue at the back of the Mental Health building.
2. The Beck Anxiety Inventory to assess the change in the participant's level of anxiety.
3. Physiological and anthropometric: Blood pressure and heart rate, body weight and height to calculate body mass index (BMI), skinfold caliper assessment to calculate percent body fat, waist and hip circumference to calculate waist to hip ratio at baseline and 60 days.
4. Physical activity: Physical activity will be assessed at baseline and 30- and 60-days follow-up by the Stanford 7-day Activity Recall. This instrument assesses the amount (number of hours) of moderate, physically challenging, and very physically challenging activities over the past 7 days. This instrument provides useful estimates of habitual physical activity for research, significantly agrees with daily self-report of physical activity, and has been validated for use in community settings.
5. Quality of life: The SF-36v2™ Health Survey provides psychometrically-based physical and mental health summary measures and a preference-based health utility index. It is a generic measure that does not target a specific age, disease, or treatment group and will be assessed at baseline and 30- and 60-days follow-up.

Participant Compensation Subjects will be compensated $40 for attending each assessment at baseline and 30- and 60-days follow-up. This amount is intended to compensate for their time and effort in completing the outcome and assessment measures. Therefore, a subject could receive up to $120 for participating in the study. We believe this amount to be fair and not to constitute coercion, given the commitment required for completing the entire protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 years and over.
* Individuals with a diagnosed type or form of depression.
* An elevated level of homocysteine (> 10 µmol/L) at screening.
* Interest in participating in a novel nutritional supplement program.
* Willingness to follow recommendations, including going off of all medication for depression 2 weeks before starting vitamin B complex regimen.

Exclusion Criteria:

* Excluded in any of the above criteria are not met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Depression level | 2 months
  Assessed by the Beck Depression Inventory II, the Beck Anxiety Inventory, SF-36v2™ Health Survey, physiological and anthropometric measures
  Because item 9 of the Beck Depression Inventory inquires about "Suicidal thoughts or wishes," we will immediately notify the attending physician in the Crisis facility of UM/JMH if a subject responds affirmatively to this question, which may be indicative of suicidal ideation (SI).

CONTACTS AND LOCATIONS:
Overall Officials: John E Lewis, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami CRB, Miami, Florida, United States